CLINICAL TRIAL: NCT05071170
Title: Satiety Responses and Oral Processing Characteristics of Commonly Consumed Meals
Acronym: EAT
Status: Completed | Type: Observational
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-036
Record Dates: First submitted 2021-09-07; First posted 2021-10-08 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Adults
Keywords: Eating behaviour; Eating rate; Texture; Satiety; Sensory
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Degree of food processing and food texture: Processed vs unprocessed foods based on NOVA classification
  Soft and hard foods manipulated by cooking method
  Interventions: Behavioral: Ad libitum energy intake

INTERVENTIONS:
Behavioral: Ad libitum energy intake — Investigate post meal satiety and subsequent post meal energy intake according to degree of food processing and eating behaviour

SUMMARY:
Rationale: Oral processing behaviours (i.e. eating rate, bite size, chews per bite, oral exposure time etc.) play a major role in food ingestion and digestion, and potentially influence satiation and satiety responses . Experimental studies showed that a prolonged mastication or a slower eating rate is associated with decreased food intake , and increased satiety response per kcal consumed. Therefore, one possible approach to control the intake and appetite is to encourage eating behaviour that slow the rate of food intake and enhance the onset of satiety. Texture led changes to oral processing behaviours could offer an exciting opportunity to adapt an individual's response to structure properties of the food being consumed in a way that maintains the associated eating experience and satiety from food intake.

However, no studies to date have investigated how differences in food processing influences food texture characteristics and oral processing behaviours, and subsequently impact on individuals' satiety responses and their subsequent food intake. The proposed study will examine the role of oral processing behaviours and/ or food processing (i.e. minimally processed, processed and ultra-processed) on satiety responses and the subsequent food intake

Objectives: The objectives of the study are to characterise the differences in oral processing behaviours (i.e. eating rate, bite size, chew per bite, oral exposure time etc.) and satiety responses of meals that differ in their degree of processing, and to further investigate how texture-based differences in oral processing behaviours modified by degree of food processing influence the satiety responses (fullness over the time) and subsequent food intake.

Study design: A total of 1 screening session (Session 1) and 4 test sessions (Sessions 2 to 5) and 2x2 randomised crossover design where participants receive 4 treatments (i.e. 4 test meals) over 4 test sessions

Study population: Healthy males ( n=50), aged 21-50 years with BMI between 18-25 kg/m2

Intervention: Session 1 involves tasting of up to 16 food items and computer task to rate and evaluate their perception and health behaviour. Sessions 2 to 5 involve evaluation of sensory characteristics, video recording of participants eating, and wrist-worn accelerometer to track wrist movement while consuming the 4 test meals.

DETAILED DESCRIPTION:
Objectives:

The objectives of the study are to characterise the differences in oral processing behaviours (i.e. eating rate, bite size, chew per bite, oral exposure time etc.) and satiety responses of meals that differ in their degree of processing, and to further investigate how texture-based differences in oral processing behaviours modified by degree of food processing (i.e. un-, minimally-processed, processed and ultra-processed foods) influence the satiety responses (fullness over the time) and subsequent food intake.

Study Design:

The current study will require participants to attend a total of 5 study sessions involving 1 screening session (session 1) and 4 test sessions (sessions 2 to 5). Each session will last for approximately one to 1.5 hours (Screening), or 1.5 to 3 hours each (4 test sessions), respectively. maximum of 50 participants will be recruited for this study.

The perceived sensory, oral processing behaviours, and satiety responses across different meals (e.g. rice with meat and vegetable, meat with potato and salad, etc.) will be assessed using video recording, sensory and appetite assessment on 100mm Visual Analogue Scale (VAS), respectively. The subsequent food intake at the ad libitum snack for different meals will also be measured using a Sartorius balance. The dietary behaviour, perception and portion selection of foods varying in level of processing and nutrient sources will also be evaluated using a Health Behaviour Questionnaire and a simple computerised task.

Test Foods:

All food that are consumed are commercially available, safe for human consumption and prepared in line with safe hygienic food preparation (e.g. Meals: rice with meat and vegetable, meat with potato and salad etc.; Sweet and savoury snacks: biscuits, chips etc.)

Screening (Session 1, 1-1.5 hour):

All potential participants will be asked to give informed consent before taking part in any of the research activities. Participants are to complete a screening questionnaire and basic anthropometric measurements such as height, weight, skinfold measurements and percentage body fat using a Bioelectrical Impedance Analyser (Tanita) will be taken.

Successfully screened participants will proceed to complete a Food Preference Questionnaire, Health Behaviour Questionnaire and taste no more than 16 samples to rate and evaluate their perception and health behaviour for the foods varying in degree of processing and nutrient sources at the remaining of the screening session.

Test sessions (Sessions 2 to 5, 1.5 to 3 hours each):

Participants will attend 1 session per week for four consecutive weeks to evaluate up to 4 fixed portion test meals across for lunch-time sessions, i.e. 1 fixed portion test meal per session. On each test day, participants will also be asked to consume 1 ad libitum snack after 2 hours of consuming the fixed portion test meal.

Participant will be required to fast from 11.00 pm the evening before and refrain from engaging in vigorous physical activities.

On each test day, participants will be asked to arrive at CNRC between 8.00-9.00am and complete a set of appetite ratings (pre-breakfast rating). Following the pre-breakfast rating, participants will receive a standardised, fixed portion breakfast to take away with them and consume at fixed interval during the morning (before the lunch). The purpose is to equilibrate their appetite need state ahead of the fixed portion test meal at lunch session. Participants will consume the breakfast within 15 minutes, after which complete a second set of appetite ratings (post-breakfast ratings). Participants will refrain from consuming anything except water and continue to complete the appetite rating at 15 or 30 minutes' intervals before coming to CNRC for their lunch (between 12.00-1.00pm), prompted by reminder set on their mobile device.

The lunch session will be scheduled from midday onwards (between 12.00-1.00pm) and will begin with a set of appetite rating (pre-lunch rating). Participants will be served a fixed portion test meal along with a glass of water. Participants will then be asked to consume the fixed portion test meal within 20 minutes. Participants' eating behaviour at lunch will be webcam recorded in order to record and behaviourally code their oral processing behaviour (i.e. eating rate, bite number, bite size etc). In addition, Participants will be asked to wear a wrist worn accelerometer (M5StickC ESP32-PICO Mini loT Development Kit, China) on the hand they eat with to track the wrist movement while eating. After completed eating, participants will be required to rate its sensory characteristics, such as liking, familiarity, overall flavour intensity, firmness, crunchiness, chewiness, saltiness and sweetness etc on a 100mm Visual Analogue Scale (VAS) using a computer. Participants will be required to complete post-lunch appetite ratings at 15 or 30 minutes' intervals for 120 minutes (post-lunch ratings).

After approximately two hours, participants will return to CNRC for an ad-libitum afternoon snack, and rate their appetite before consuming the ad-libitum snack. Participants will be instructed to consume in their normal way and to eat until comfortably full. Participants will leave CNRC after the snack session and asked to complete a food diary to record his food intake for the rest of the day.

The sensory, oral processing characteristics, and satiety responses for 4 different fixed portion test meals will be assessed. The subsequent food intake at ad libitum snack for different meals will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male
* Aged between 21 and 50-year-old
* Are of normal weight (BMI 18-25kg/m2)
* Stable weight for the previous 12 months (<5kg weight fluctuation in the previous year)
* Healthy dentition and ability to bite, chew and swallow normally
* No history of pain or discomfort in jaw movements or excessive teeth clenching or grinding
* No caries or periodontal disease

Exclusion Criteria:

* Are a smoker
* Have any dislikes, intolerances or allergies to foods or common food ingredients e.g. nuts, soya, wheat, gluten, cereal, fruits, biscuits, dairy products, rice, vegetable, meat, seafood, sugar and sweetener, gelatin, natural food colourings or flavourings (e.g. MSG), etc.
* Have any specific dietary requirements and/ or restrictions (e.g. Vegan/ vegetarian, religious beliefs, lactose intolerance, calorie restricted diet etc.)
* Have sinus problems that affect your taste and smell
* Have known glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Are taking insulin or medication known to affect your appetite or metabolism
* Have major chronic diseases such as heart disease, cancer or diabetes mellitus
* Have active Tuberculosis (TB) or currently receiving treatment for TB
* Have any known Chronic Infection or known to suffer from or have previously suffered from or is a carrier of Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV)
* Are a member of the research team or their immediate family members. Immediate family member is defined as a spouse, parent, child, or sibling, whether biological or legally adopted
* Are enrolled in a concurrent research study judged not to be scientifically or medically compatible with the study of the CNRC

Ages: 21 Years to 50 Years | Sex: Male
Age Groups: Adult
Study Population: Study population will be recruited from the National University of Singapore via advertisements posted in public notice boards at the campus, local food shops and cafes, and approved websites.Potential study participants will also be recruited from existing database of previous study participants who have provided permission to be contacted for participants in future research projects. Word of mouth and email will also be used to recruit potential participants.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Oral processing behaviour | During test session 2, Up to 20 minutes
  Participants will be video-recorded during the lunch sessions to measure oral processing behaviour (e.g., derived from number of bites, chews, swallows and eating duration) of the test fixed portion test meals using an annotation software.
Oral processing behaviour | During test session 3, Up to 20 minutes
  Participants will be video-recorded during the lunch sessions to measure oral processing behaviour (e.g., derived from number of bites, chews, swallows and eating duration) of the test fixed portion test meals using an annotation software.
Oral processing behaviour | During test session 4, Up to 20 minutes
  Participants will be video-recorded during the lunch sessions to measure oral processing behaviour (e.g., derived from number of bites, chews, swallows and eating duration) of the test fixed portion test meals using an annotation software.
Oral processing behaviour | During test session 5, Up to 20 minutes
  Participants will be video-recorded during the lunch sessions to measure oral processing behaviour (e.g., derived from number of bites, chews, swallows and eating duration) of the test fixed portion test meals using an annotation software.
Change in Post breakfast satiety responses | During test session 2, at 15 or 30 minutes' intervals, up to 4 hours each
  Participants will be asked rate their appetite sensations using a visual analogue scale (VAS) pre- and post meals. VAS is anchored at 'Not at all' (0) to 'Extremely' (100), where a higher score will indicate greater intensity.
Change in Post breakfast satiety responses | During test session 3, at 15 or 30 minutes' intervals, up to 4 hours each
  Participants will be asked rate their appetite sensations using a visual analogue scale (VAS) pre- and post meals. VAS is anchored at 'Not at all' (0) to 'Extremely' (100), where a higher score will indicate greater intensity.
Change in Post breakfast satiety responses | During test session 4, at 15 or 30 minutes' intervals, up to 4 hours each
  Participants will be asked rate their appetite sensations using a visual analogue scale (VAS) pre- and post meals. VAS is anchored at 'Not at all' (0) to 'Extremely' (100), where a higher score will indicate greater intensity.
Change in Post breakfast satiety responses | During test session 5, at 15 or 30 minutes' intervals, up to 4 hours each
  Participants will be asked rate their appetite sensations using a visual analogue scale (VAS) pre- and post meals. VAS is anchored at 'Not at all' (0) to 'Extremely' (100), where a higher score will indicate greater intensity.
Change in Post lunch satiety responses | During test session 2, 15 or 30 minutes' intervals, up to 2 hours each
  Participants will be asked rate their appetite sensations using a visual analogue scale (VAS) pre- and post meals. VAS is anchored at 'Not at all' (0) to 'Extremely' (100), where a higher score will indicate greater intensity.
Change in Post lunch satiety responses | During test session 3, 15 or 30 minutes' intervals, up to 2 hours each
  Participants will be asked rate their appetite sensations using a visual analogue scale (VAS) pre- and post meals. VAS is anchored at 'Not at all' (0) to 'Extremely' (100), where a higher score will indicate greater intensity.
Change in Post lunch satiety responses | During test session 4, 15 or 30 minutes' intervals, up to 2 hours each
  Participants will be asked rate their appetite sensations using a visual analogue scale (VAS) pre- and post meals. VAS is anchored at 'Not at all' (0) to 'Extremely' (100), where a higher score will indicate greater intensity.
Change in Post lunch satiety responses Session 5 | During test session 5, 15 or 30 minutes' intervals, up to 2 hours each
  Participants will be asked rate their appetite sensations using a visual analogue scale (VAS) pre- and post meals. VAS is anchored at 'Not at all' (0) to 'Extremely' (100), where a higher score will indicate greater intensity.
Subsequent food intake post test meal | During test session 2, up to 0000hrs
  Participants will be asked to bring a food dairy home to record their food and beverage intake for the rest of the test day. This is to assess participants' calorie intake for the remaining day on the test session.
Subsequent food intake post test meal | During test session 3, up to 0000hrs
  Participants will be asked to bring a food dairy home to record their food and beverage intake for the rest of the test day. This is to assess participants' calorie intake for the remaining day on the test session.
Subsequent food intake post test meal | During test session 4, up to 0000hrs
  Participants will be asked to bring a food dairy home to record their food and beverage intake for the rest of the test day. This is to assess participants' calorie intake for the remaining day on the test session.
Subsequent food intake post test meal | During test session 5, up to 0000hrs
  Participants will be asked to bring a food dairy home to record their food and beverage intake for the rest of the test day. This is to assess participants' calorie intake for the remaining day on the test session.

CONTACTS AND LOCATIONS:
Overall Officials: Pey Sze Teo, PhD, Principal Investigator — Singapore Institute Of Food and Biotechnology Innovation (SIFBI), A*STAR
Locations (1):
- Singapore Institute of Food and Biotechnology Innovation (SIFBI)/Clinical Nutrition Research Centre, Singapore, Singapore